CLINICAL TRIAL: NCT05145270
Title: A Comparative Study on Efficacy and Safety of add-on Sulforaphane or rTMS to Escitalopram for Major Depressive Disorder With Poor Response to Initial Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHDC12019X09
Record Dates: First submitted 2021-12-02; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Sulforaphane; rTMS; Efficacy; Oxidative stress; Marker; Add-on
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Intervention Model Description: All the participants will be 1:2:2 randomly assigned to different intervention groups including escitalopram, escitalopram plus sulforaphane (SFN) , and escitalopram plus repetitive transcranial magnetic stimulation (rTMS).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Escitalopram (Active Comparator): The dose of Escitalopram based on treatment guidelines for major depressive disorder and drug prescription manual is 10-20mg/day, once per day.
  Interventions: Drug: Escitalopram
- Escitalopram plus Sulforaphane (Experimental): The dose of Escitalopram based on treatment guidelines for major depressive disorder and drug prescription manual is 10-20mg/day, once per day.
  The oral dose of SFN is based on weight. The usage and dosage are as follows: 40-70kg, 4 tablets/day (containing 274μmol of glucosinolates); 70-90kg, 6 tablets/day (containing 411μmol of glucosinolates). Take it once in the morning and evening.
  Interventions: Dietary Supplement: Escitalopram+Sulforaphane; Drug: Escitalopram
- Escitalopram plus rTMS (Experimental): The dose of Escitalopram based on treatment guidelines for major depressive disorder and drug prescription manual is 10-20mg/day, once per day.
  rTMS is delivered to the left dorsolateral prefrontal lobe position. Stimulation parameters are set to be 80 stimulation strings of 10Hz with an interval of 12 seconds. Each stimulation string includes 30 stimulations lasting for 3 seconds. One session includes 2400 stimulation strings lasting for 19 minutes and 40 seconds. The course of rTMS treatment includes 20 sessions, once a day or twice a day.
  Interventions: Device: Escitalopram+rTMS; Drug: Escitalopram

INTERVENTIONS:
Dietary Supplement: Escitalopram+Sulforaphane — Escitalopram(No-specified) 10-20mg/d, once per day; Sulforaphane(ZHIYINGUOSU, Shenzhen Fushan Biotech Co. Ltd.). 40-70kg, 4 tablets/day (containing 274μmol of glucosinolates); 70-90kg, 6 tablets/day .
  Arms: Escitalopram plus Sulforaphane
Device: Escitalopram+rTMS — Escitalopram(No-specified) 10-20mg/d, once per day; rTMS: rTMS is delivered to the left dorsolateral prefrontal lobe position. Stimulation parameters are set to be 80 stimulation strings of 10Hz with an interval of 12 seconds. Each stimulation string includes 30 stimulations lasting for 3 seconds. One session includes 2400 stimulation strings lasting for 19 minutes and 40 seconds. The course of rTMS treatment includes 20 sessions, once a day or twice a day.
  Arms: Escitalopram plus rTMS
Drug: Escitalopram — Escitalopram(No-specified) 10-20mg/d, once per day.

SUMMARY:
A 12-week, randomized controlled trial (RCT) with parallel grouping design will be conducted to compare the efficacy and safety of different treatments. One hundred and eighty adults diagnosed with major depressive disorder (MDD) with no or poor response to initial antidepressant treatment will be recruited. Then all the patients will be 1:2:2 randomly assigned to different intervention groups including escitalopram, escitalopram plus sulforaphane (SFN) , and escitalopram plus repetitive transcranial magnetic stimulation (rTMS). Clinical symptoms and side-effects will be evaluated or recorded using the 17-Hamilton Depression Rating Scale (17-HDRS), the Hamilton Anxiety Scale (HAMA), side-effects sheet, etc., at Critical Decision Points (CDP) including weeks 2, 4, 8 and 12 after treatment. Blood cell counting, biochemical, and electrocardiogram examination will be performed at weeks 4, 8 and 12 after treatment in order to evaluate the effect of different interventions on the physical condition. In addition, niacin skin flush response and serum markers including nuclear factor erythroid-2-related factor 2(Nrf-2), p-Nrf2, malondialdehyde (MDA), superoxide dismutase (SOD) and erythrocyte glutathion peroxidase (GPX) will be tested at baseline and endpoint. The primary outcome is the reduction rate in 17-HDRS total score from baseline to the end of the study. The secondary outcomes include changes in niacin skin flush response test and levels of serum markers. All the data will be analyzed by SPSS software.

ELIGIBILITY:
The inclusion criteria are as follows:

1. aged 18-60 years;
2. diagnosed with moderate or severe depressive disorder according to the criteria of the DSM-5;
3. total score of 17-HDRS≥17;
4. never receiving electroconvulsive therapy (ECT)/modified ECT (MECT)/rTMS or other treatments in the past month;
5. no response or poor response (having a reduction of <20% on the total score of the 17-item Hamilton Depression Scale compared with the baseline) to adequate antidepressants (except escitalopram) treatment for at least 4 weeks;
6. having sufficient audio-visual ability and comprehension;
7. signed informed consent statements.

The exclusion criteria are as follows:

1. serious or active somatic illness (abnormal index values were more than twice the limit of normal);
2. a history of mania/hypomania;
3. current high risk of suicide (score of item 3 of 17-HDRS ≥ 3);
4. pregnant or lactating women, or planning pregnant women;
5. taking immunosuppressants or vitamins recently.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
the reduction rate in 17-HDRS total score from baseline to the end of the study | at baseline, week 2/4/8/12 after treatment.
  Remission is defined as 17-HDRS total score ≤7; Response is defined as ≥50% decrease from 17-HDRS total score at baseline and 17-HDRS total score>7; Nonresponse is defined as having a reduction of<50% on the total score of 17-HDRS comparing with baseline.

SECONDARY OUTCOMES:
changes in levels of serum markers from baseline to the end of the study | at baseline, week 8-12 after treatment.
  changes in levels of serum markers including nuclear factor erythroid-2-related factor 2(Nrf-2), p-Nrf2, malondialdehyde (MDA), superoxide dismutase (SOD) and erythrocyte glutathion peroxidase (GPX)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided